CLINICAL TRIAL: NCT04933578
Title: Children and Parents' Preferences About the Appearance of Dentists With Respect to Personal Protective Equipment in Pediatric Dentistry
Brief Title: Preferences About Personal Protective Equipment
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sema Aydınoglu, assistant professor, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 81
Record Dates: First submitted 2021-06-18; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Dental Anxiety; Behavior, Child; Preference, Patient
Keywords: Personal protective equipment; dental anxiety; parents; preferences; health care professionals
MeSH Terms: conditions — Child Behavior; Patient Preference

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children: 1. The Faces Version of Modified Child Dental Anxiety Scale (MCDASf), which is a psychometric dental anxiety scale for children with eight questions, was used to determine the dental anxiety levels of the children.
  2. The children's preferences for the appearance of dentists were determined in the second part.
  3. Routine dental examinations of children with a dental mirror and artificial light were completed by an experienced pediatric dentist according to the World Health Organization (WHO) guidelines and criteria.
  Interventions: Behavioral: Dental anxiety scales
- Parents: 1. The questionnaire including demographic information (age, sex, and medical and dental history) was applied to the parents.
  2. In the second section, the MDAS was administered to parents, differently from children.
  3. The parents' preferences for the appearance of dentists were determined in the second part.
  Interventions: Behavioral: Dental anxiety scales

INTERVENTIONS:
Behavioral: Dental anxiety scales — * The Faces Version of Modified Child Dental Anxiety Scale (MCDASf), which is a psychometric dental anxiety scale for children with eight questions, was used to determine the dental anxiety levels of the children. The scores of each question are represented by varying cartoon faces according to emotions ranging from 1 'relaxed' to 5 'very anxious'. The total scores range from 8 to 40. The scores were categorized as not anxious (>9), slightly anxious (9-16), fairly anxious (17-24), very anxious (25-32), and extremely anxious (33-40).
  * the Modified Dental Anxiety Scale (MDAS) was administered to parents, differently from children. The MDAS has five questions. The scores of each question range from 1 'relaxed' to 5 'very anxious.' The total score ranges from 5 to 25.

SUMMARY:
Personal protective equipment (PPE) gained importance during the Coronavirus Disease 2019 (COVID-19) pandemic, which is a global hot topic for all healthcare staff.

DETAILED DESCRIPTION:
To assess children and parents preferences about dentists' appearance concerning their PPE and to determine the relationship between the preferences of the children and their parents.

A total of 250 children aged with 6-12 years and their parents were enrolled in the study. Standardised pictures with different sex, attire, eye protector, hair protector, mask and gloves were shown to children and their parents separately and asked to chose their preferences. Dental anxiety of children and their parents were determined with MCDASf and MDAS, respectively. Decayed-missing-filled teeth (DMFT) index was employed to the children.

ELIGIBILITY:
Inclusion Criteria:

* aged 6-12 years and their parents,
* intellectually sufficient to complete the questionnaire,
* with voluntariness to take part in the study

Exclusion Criteria:

* had mental or physical disorders, cooperation problems or dental pain

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children who presented for the first time to the Faculty of Dentistry in Rize and their parents
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
To assess children and parents preferences about dentists' appearance concerning their PPE and to determine the relationship between the preferences of the children and their parents according to dental anxiety levels. | for two months from the beginning of the study
  Standardised pictures with different sex, attire, eye protector, hair protector, mask and gloves were shown to children and their parents separately and asked to chose their preferences. Dental anxiety of children and their parents were determined with MCDASf and MDAS, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Sema Aydinoğlu, Rize, Turkey (Türkiye)